CLINICAL TRIAL: NCT06595966
Title: Exploratory Research on Constructing a Computational Biological Model Based on Next Generation Sequencing Technology for Monitoring Measurable Residual Disease (MRD) After Breast Cancer Surgery
Brief Title: Exploratory Research on Constructing a Computational Biological Model Based on NGS for MRD After Breast Cancer Surgery
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-0693
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer; Measurable Residual Disease
MeSH Terms: conditions — Breast Neoplasms; Neoplasm, Residual

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- experimental group: The results of CA15-3, CEA, color Doppler ultrasound and other traditional postoperative monitoring examinations for breast cancer, as well as 5ml of peripheral venous blood, were collected on the day of enrollment/the 7th day after adjuvant treatment/the 3rd, 6th, 9th, 12th, 15th, 18th, 21st, 24th, 30th and 36th months after surgery.

SUMMARY:
This study will include 80 subjects after radical breast cancer resection, collect blood samples of the above subjects, observe and quantify the characteristic changes of cfDNA in the blood of breast cancer subjects after surgery, and establish a computational biological model based on next generation sequencing to monitor breast cancer MRD;

DETAILED DESCRIPTION:
This study will include 80 subjects after radical breast cancer resection. The results of CA15-3, CEA, color Doppler ultrasound and other traditional postoperative monitoring examinations for breast cancer, as well as 5ml of peripheral venous blood, were collected on the day of enrollment/the 7th day after adjuvant treatment/the 3rd, 6th, 9th, 12th, 15th, 18th, 21st, 24th, 30th and 36th months after surgery. We observe and quantify the characteristic changes of cfDNA in the blood of breast cancer subjects after surgery, and establish a computational biological model based on next generation sequencing to monitor breast cancer MRD;

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥ 18 years old, gender not limited; 2. Obtain plasma samples from the subjects during a 3-year follow-up period; 3. The subjects fully understand the study and voluntarily sign the informed consent form; 4. Able to cooperate with a 3-year follow-up visit to the hospital; 5. The physical fitness status score (ZPS) of the ECOG scoring criteria for the subjects must be ≤ 1; 6. Life expectancy ≥ 5 years; 7. Subjects who meet the following criteria:

  1. Histopathology confirmed primary breast cancer (unlimited molecular type);
  2. Radical breast cancer resection is expected;
  3. Adopting postoperative adjuvant therapy or preoperative neoadjuvant therapy;

Exclusion Criteria:

* 1. The subject is pregnant or breastfeeding; 2. Serious mental illness or drug abuse; 3. Unable to obtain the subject's plasma during this period; 4. If the subject has a non primary malignant tumor of the breast with a clear pathological diagnosis within 5 years before enrollment: 5. If the subject has suspected non breast malignant tumors (such as B-ultrasound, CT, etc.) on imaging within the past year of enrollment, but without pathological confirmation; 6. Clinical suspicion of distant metastatic lesions; 7. The subject has received any blood product infusion therapy within the past 30 days; 8. Known carriers of pathogenic genetic mutations;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eighty patients with breast cancer were diagnosed in the Second Affiliated Hospital of Zhejiang University School of Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Sample Sizes | 3 years
  The number of samples that meet the requirements meets the statistical requirements

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

DOCUMENTS (2):
  • Study Protocol (2023-06-07): https://cdn.clinicaltrials.gov/large-docs/66/NCT06595966/Prot_000.pdf
  • Informed Consent Form (2023-06-07): https://cdn.clinicaltrials.gov/large-docs/66/NCT06595966/ICF_001.pdf